CLINICAL TRIAL: NCT05064891
Title: Application of Ultrasound Imaging of Suprascapular Nerves and Dynamic Shoulder Movement for Stroke Patients
Brief Title: Ultrasound Application on the Suprascapular Nerve and Dynamic Shoulder Movement for Stroke Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202104006RIND
Record Dates: First submitted 2021-09-09; First posted 2021-10-01 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-06

CONDITIONS: Stroke
Keywords: Ultrasonography; Stroke; Suprascapular Nerve; Pain
MeSH Terms: conditions — Stroke; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke patients
  Interventions: Procedure: Ultrasound guided injection
- Participants without stroke

INTERVENTIONS:
Procedure: Ultrasound guided injection — Subdeltoid bursa injection, suprascapular nerve block, or posterior glenohumeral joint injection. The participants should only receive one type of the injection mentioned above.
  Groups: Stroke patients

SUMMARY:
The suprascapular nerve is the first nerve that branches from the upper trunk of brachial plexus. It receives signals transmitted from the fifth and sixth cervical root. The clinical importance of suprascapular nerve is mainly based on its distribution of 70% sensory innervation to the glenohumeral joint. After being divided from the upper trunk, the suprascapular nerve goes laterally and posteriorly. First, it passes underneath the omohyoid muscle, and then goes through the suprascapular notch into the suprascapular fossa. If there are some problems inside the supraspinatus muscle at the suprascapular fossa, the suprascapular nerve below it may be compromised. After the suprascapular nerve passes the suprascapular fossa, it courses through the spinoglenoid notch, and then goes into the infraspinatus fossa to innervate the infraspinatus muscle. Based on the sensory and motor innervation of the suprascapular nerve to the shoulder joint, the sonographic images of the suprascapular nerves would add tremendous values in assessing patients with refractory shoulder pain. Although there are some studies trying to measure the size of the suprascapular nerve, no available research can be found in stroke patients. Our study aims to explore the ultrasound morphology of the suprascapular nerves as well as subacromial dynamic imaging in patients with stroke. A control group without stroke will be recruited for comparison.

DETAILED DESCRIPTION:
Introduction:

Shoulder pain arises to be one of the most common musculoskeletal complaints, and with the high prevalence in stroke patients. The mechanism of an increased risk of painful shoulders is multifactorial and the role of the suprascapular nerve in development and management of shoulder pain has been highlighted recently. In recent years, high resolution ultrasound has been widely applied on evaluation of entrapment neuropathy, and its reliability on assessing the cross-sectional area of supraspcapular nerves has been validated. As the suprascapular nerve is crucial for conducting shoulder motion and sensation, it is of clinical importance to measure the size of suprascapular nerve. Our study aims to explore the ultrasound morphology of the suprascapular nerves as well as subacromial dynamic imaging in patients with stroke and to investigate the nerve's size after ultrasound-guided injection.

Material and methods:

Participants: Adult stroke patients (≥ 20 year old).

Control: Asymptomatic adult subjects (≥20 year old)

Exclusion criteria:

The exclusion criteria included history of malignancy, uncontrolled medical conditions (like systemic rheumatic disease, including rheumatic arthritis and ankylosing spondylitis), previous major trauma or surgeries, suprascapular nerve block on either side of the shoulders within the three months, and the patients with specific aphasia and poor cognition.

Study design:

This was a longitudinal follow-up study investigating the suprascapular nerves, the dynamic subacromial examination of shoulder, and the nerve's size after ultrasound-guided injection in patients with stroke. All the participants were required to ambulate independently, have normal cognitive function and complete the given questionnaires. The study included at least 60 participants.

Detail of the investigation

1. High-resolution ultrasound evaluation of the shoulder region was applied to recognize the biceps tendon, subscapularis tendon, supraspinatus tendon, and infraspinatus tendon.
2. High-resolution ultrasound evaluation was applied for the C5, C6 and C7 nerve roots and the suprascapular nerve over the supraclavicular fossa, in the supraspinatus fossa and in the infraspinatus fossa to obtain the nerve cross-sectional image.
3. High-resolution ultrasound evaluation was applied for the dynamic examination of the shoulder to recognize the impingement of the shoulder.
4. The investigators collected the shoulder pain-related information, including physical examination results (bicipital groove tenderness, Speed test, Yergason's test, Empty can test, Neer test, Hawkins-Kennedy test and painful arc test) and status of disability using Shoulder Pain and Disability Index (SPADI).
5. The investigators collected the information of the types of the stroke, onset times, and functional status, including Bathel index and Fugl-Meyer Upper Extremity Assessment.

Outcome measurement:

Primary outcome:

1. The measurements of the nerve cross-sectional area were conducted by another specialist with the image processing software (Image J). For the most proximal section of the suprascapular nerve, the cross-section of the nerve fascicles inside the hyperechoic epineurium were measured. In the segment over the supraspinatus and infraspinatus fossae, the whole nerve's cross-section including its epineurium were measured. The data collection was performed at the initial recruitment and one month later after the injection.
2. The Chinese version of the Shoulder Pain and Disability Index (SPADI) tool. The data collection was performed at the initial recruitment and one month later after the injection.
3. Visual analogue scale. The data collection was performed at the initial recruitment and one month later after the injection.
4. The range of the motion and impingement of the shoulder under dynamic subacromial examination. The data collection was performed at the initial recruitment and one month later after the injection.

Statistical analysis:

1. Continuous variables: Mann Whitney u test
2. Categorical variables: Chi-square test

ELIGIBILITY:
Inclusion Criteria:

* Adult and stroke patients (≥ 20 year old). All the participants were those visiting the department of physical medicine and rehabilitation for musculoskeletal complaints.

Exclusion Criteria:

* History of malignancy
* Uncontrolled medical conditions (like systemic rheumatic disease, including rheumatic arthritis and ankylosing spondylitis).
* Previous major trauma or surgeries, and suprascapular nerve block on either side of the shoulders within the three months.
* The patients with specific aphasia and poor cognition.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult and stroke patients (≥ 20 year old). All the participants were those visiting the department of physical medicine and rehabilitation for musculoskeletal complaints.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Nerve cross-sectional area at the recruited time | at the recruited time
  The measurements of the nerve cross-sectional area were conducted by another specialist with the image processing software (Image J). For the most proximal section of the suprascapular nerve, the cross-section of the nerve fascicles inside the hyperechoic epineurium were measured. In the segment over the supraspinatus and infraspinatus fossae, the whole nerve's cross-section including its epineurium were measured.
Change from the baseline of nerve cross-sectional area after the injection | at one month later after the injection
  The measurements of the nerve cross-sectional area were conducted by another specialist with the image processing software (Image J). For the most proximal section of the suprascapular nerve, the cross-section of the nerve fascicles inside the hyperechoic epineurium were measured. In the segment over the supraspinatus and infraspinatus fossae, the whole nerve's cross-section including its epineurium were measured.
Dynamic shoulder motion under ultrasound imaging | Baseline and after intervention (if available)
  Subacromial motion metrics, based on the reciprocol movement of the greater tubercle of the humerus in relation to the acromion
The Chinese version of the Shoulder Pain and Disability Index at the recruited time | at the recruited time
  The Chinese version of the Shoulder Pain and Disability Index (SPADI) tool. The SPADI tool consisted of 13 questions categorized in two domains: pain and disability. They were instructed to indicate the level of influence on a 10 cm visual analogue scale for each question with a rating from 0 (no pain or no difficulty) to 10 (worst pain or extreme difficulty). The scores from the pain and functional domains were averaged to generate the total score of SPADI, with a highest value of 100 points.
Change from the baseline of The Chinese version of the Shoulder Pain and Disability Index at recruited time after the injection | at one month later after the injection
  The Chinese version of the Shoulder Pain and Disability Index (SPADI) tool. The SPADI tool consisted of 13 questions categorized in two domains: pain and disability. They were instructed to indicate the level of influence on a 10 cm visual analogue scale for each question with a rating from 0 (no pain or no difficulty) to 10 (worst pain or extreme difficulty). The scores from the pain and functional domains were averaged to generate the total score of SPADI, with a highest value of 100 points.
Visual analogue scale at the recruited time | at the recruited time
  The pain scale to evaluate pain, from 0 to 10. The lower means less pain.
Change from the baseline of Visual analogue scale after the injection | at one month later after the injection
  The pain scale to evaluate pain, from 0 to 10. The lower means less pain.
Range of the motion and impingement at the recruited time | at the recruited time
  Range of the motion of the shoulder, from 0 degree to 180 degree. The lower means more limitation. The impingement of supraspinatus tendon, subdeltoid bursa and acromion are evaluated under ultrasonography. The transducer is positioned along the scapular plane lateral to the acromion. The participant gradually raises the arm, and the examiner simultaneously observes whether there is bulging of the subacromial bursa and abnormal elevation/movement of the humeral head.
Change from the baseline of range of the motion and impingement after the injection | at one month later after the injection
  Range of the motion of the shoulder, from 0 degree to 180 degree. The lower means more limitation. The impingement of supraspinatus tendon, subdeltoid bursa and acromion are evaluated under ultrasonography. The transducer is positioned along the scapular plane lateral to the acromion. The participant gradually raises the arm, and the examiner simultaneously observes whether there is bulging of the subacromial bursa and abnormal elevation/movement of the humeral head.

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Vin Chang, MD,PhD, Study Chair — National Taiwan University Hospital Bei-Hu Branch
Locations (1):
- National Taiwan University Hospital, Bei-Hu Branch, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu CH, Chang KV, Ozcakar L, Hsiao MY, Hung CY, Shyu SG, Wang TG, Chen WS. Sonographic tracking of the upper limb peripheral nerves: a pictorial essay and video demonstration. Am J Phys Med Rehabil. 2015 Sep;94(9):740-7. doi: 10.1097/PHM.0000000000000344. PMID 26135374
- [Result] Chang KV, Hung CY, Wang TG, Yang RS, Sun WZ, Lin CP. Ultrasound-Guided Proximal Suprascapular Nerve Block With Radiofrequency Lesioning for Patients With Malignancy-Associated Recalcitrant Shoulder Pain. J Ultrasound Med. 2015 Nov;34(11):2099-105. doi: 10.7863/ultra.14.12042. Epub 2015 Oct 9. PMID 26453125
- [Result] Chang KV, Hung CY, Wu WT, Han DS, Yang RS, Lin CP. Comparison of the Effectiveness of Suprascapular Nerve Block With Physical Therapy, Placebo, and Intra-Articular Injection in Management of Chronic Shoulder Pain: A Meta-Analysis of Randomized Controlled Trials. Arch Phys Med Rehabil. 2016 Aug;97(8):1366-80. doi: 10.1016/j.apmr.2015.11.009. Epub 2015 Dec 14. PMID 26701762
- [Result] Chang KV, Wu WT, Hung CY, Han DS, Yang RS, Chang CH, Lin CP. Comparative Effectiveness of Suprascapular Nerve Block in the Relief of Acute Post-Operative Shoulder Pain: A Systematic Review and Meta-analysis. Pain Physician. 2016 Sep-Oct;19(7):445-56. PMID 27676661